CLINICAL TRIAL: NCT00983788
Title: Evaluation of the Effect of Bezafibrate on Muscle Metabolism During Exercise in Patients With CPTII and VLCAD Deficiency
Brief Title: Effect of Bezafibrate on Muscle Metabolism in Patients With Fatty Acid Oxidation Defects
Acronym: Bezafibrate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Groupe Hospitalier Pitie-Salpetriere (Other)
Responsible Party: Principal Investigator, Mette Cathrine Oerngreen, MD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EudraCT: 2008-006704-27
Record Dates: First submitted 2009-09-23; First posted 2009-09-24 (Estimated); Last update posted 2012-05-30 (Estimated); Status verified 2012-05

CONDITIONS: Carnitine Palmitoyltransferase II Deficiency; Very Long Chain Acyl Coa Dehydrogenase Deficiency
Keywords: CPT II; VLCAD
MeSH Terms: conditions — Carnitine palmitoyl transferase 2 deficiency; VLCAD deficiency | interventions — Bezafibrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bezafibrate (Experimental)
  Interventions: Drug: Bezafibrate
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Bezafibrate — 3 x 200 mg/ day
  Arms: Bezafibrate
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The investigators propose to evaluate the effect of bezafibrate on metabolism during exercise in 22 adult patients affected with carnitine palmitoyltransferase II (CPTII) or very-long chain acyl-CoA-dehydrogenase (VLCAD) deficiencies. This study will be an 9-month, randomized, double-blind, placebo-controlled crossover trial. The trial will be conducted in two centers: Institut de Myologie, Pitié-Salpêtrière Hospital in France, and Rigshospitalet, University of Copenhagen, in Denmark. The main criteria for assessing the potential effect of this drug will be the fat oxidation rate studied during a moderate workload on cycle ergometer, after infusion of stable isotopes (palmitate and glucose tracers).

DETAILED DESCRIPTION:
Background and research aim:

Carnitine palmitoyltransferase II (CPTII) and very-long chain acyl-CoA-dehydrogenase (VLCAD) deficiencies are the two most common inherited disorders of mitochondrial fatty acid oxidation (FAO) in adults, both inherited in an autosomal recessive manner. Mitochondrial FAO plays a pivotal role for maintaining energy homeostasis in situations such as fasting, fever or prolonged exercise that require both glucose sparing and major energy supply. In these situations, a number of tissues such as skeletal muscle, heart, and liver, favour fatty acids as the main source of energy. Long-chain fatty acids (LCFA), that represent the major part of endogenous free fatty acids cannot enter the mitochondrial matrix compartment by simple diffusion, and the transfer of LCFA across the mitochondrial membranes is governed by a multienzymatic system named carnitine palmitoyltransferase (CPT) consisting of two enzymes: CPT I and II. CPT I, a key regulatory step of LCFA oxidation, is located within the outer mitochondrial membrane, while CPT II is appended to the inner face of the inner mitochondrial membrane. CPTs I and II catalyze a single reaction (carnitine + acyl-CoA ⇔ acylcarnitine + CoA~SH) in the forward and reverse directions, respectively. VLCAD is bound to the inner mitochondrial membrane, and catalyses the first step of the long-chain fatty acid β-oxidation spiral (Izai et al., 1992).

Various phenotypes of CPT II and VLACD deficiencies have been described. Severe neonatal or infantile clinical life-threatening symptoms may occur with hypoketotic hypoglycemia, liver failure, and cardiomyopathy during the first months or years of life (Demaugre et al, 1991; Bonnefont et al, 1996; Vianey-Saban et al. 1998; Andresen et al., 1999). Conversely, the "adult" forms of these diseases are more prevalent and have a clinical expression restricted to skeletal muscle. In the latter form, onset most often occurs in teenagers or young adults, and is mainly characterized by recurrent episodes of rhabdomyolysis triggered by prolonged exercise, fasting, cold or fever (DiMauro et al., 1973; Vianey-Saban et al. 1998). The major potential complication is acute renal failure following attacks of rhabdomyolysis.

Studies of fuel utilization in subjects with CPT II and VLCAD deficiencies, with stable isotopes during exercise, have shown that in vivo oxidation of LCFA was severely impaired during prolonged, low-intensity exercise. These findings indicated that residual CPT II and VLCAD activities are sufficient to maintain normal oxidation of fat at rest, but that fat oxidation rate cannot increase above basal level during exercise (Ørngreen et al., 2004; 2005).

Current recommended treatments for long-chain FAO disorders essentially relies on dietary approaches, with restriction of long-chain fat intake along with medium-chain triglyceride supply (MCT oil). A carbohydrate-rich diet also improved exercise tolerance in CPT II-deficient patients, as indicated by lowering of perceived exertion and an increased duration of exercise after such a diet (Ørngreen et al., 2003). More recently, a remarkable improvement of cardiac and muscular symptoms occurred in three children with VLCAD deficiency, after dietary supplementation with a seven-carbon medium chain fatty acid (triheptanoïn). The mechanism underlying this effect is believed to involve the production of C5 ketone bodies and propionyl-CoA, which allows for replenishment of the pool of catalytic intermediates for the citric acid cycle (Roe et al., 2002). This promising approach is still under evaluation and marked digestive side effects could restrict its indication towards the more severe form of FAO defects. Pharmacological approaches are mainly carnitine supplementation in order to provide carnitine to convert potentially toxic long-chain acyl-CoAs to acylcarnitines. However, the role of carnitine supplements in FAO defects remains controversial and of unproven value due to the absence of controlled trials.

PPARα receptors were identified as potential targets for pharmacological therapy of CPTII and VLCAD deficiencies. PPARα is a transcription factor, belonging to the superfamily of steroid-thyroid hormone receptors, which is able to modify CPT2 and VLCAD gene expression (Lemberger et al, 1996). Djouadi et al. established that administration to control mice of a CPT I inhibitor (etomoxir) causes a feedback induction of PPARα target genes involved in fatty acid oxidation such as medium-chain acyl-CoA dehydrogenase and acyl-CoA oxidase genes (Djouadi et al, 1998). PPARα was also shown to regulate the constitutive expression of the CPT2 gene and protein in the adult mouse heart and liver and to mediate up-regulation of CPT2 gene in response to fibrates in mouse liver (Aoyama et al, 1998, Watanabe et al, 2000). In humans, the "fibrate" class of hypolipidaemic drugs (clofibrate, bezafibrate, gemfibrozil, etc…) are specific ligands of PPARα and the interaction with PPARα forms the molecular basis of therapeutic effects of these drugs (Vamecq et al, 1999). The research group of Bastin J and Djouadi F hypothesized that the hypolipidemic drug bezafibrate, acting as an activator of PPARα, might stimulate FAO in CPT II and VLCAD-deficient cell lines. Bezafibrate treatment of fibroblasts from four CPT II-deficient patients with the "adult" form of the disease was shown 1) to increase the amount of CPT2 mRNA (+ 47 % to + 66 %) and the residual CPT II enzyme activity (+ 54 % to + 135 %) in a time- and dose-dependant manner, and 2) to normalize 3H-palmitate and 3H-myristate oxidation rates. Conversely, bezafibrate did not correct FAO in two patients with the "infantile" form of CPTII deficiency (Djouadi et al, 2003). Since the clinical expression of the "adult" form of CPT2 deficiency is restricted to skeletal muscle, the effect of fibrates was tested on FAO in muscle samples from such patients. After being provided with muscle samples from patients with the "adult" form of CPTII deficiency followed at the Institute of Myology (P. Laforêt, B. Eymard), it has been shown that myoblasts from these biopsies exhibited a 40 % decrease in FAO compared to control cells (Djouadi et al, 2003). Moreover, pretreatment of CPTII-deficient myoblasts with bezafibrate restored FAO to normal levels (Bastin et al, 2003).

More recently, Djouadi et al. (2005) demonstrated that addition of bezafibrate in the culture medium induced a dose-dependent (up to 3-fold) increase in palmitate oxidation capacities in fibroblasts from patients with the myopathic form of VLCAD deficiency, but not from severely affected patients. This biological improvement was related to drug-induced increases in VLCAD mRNA (+ 44 to + 150%), protein (1.5-2-fold) and residual enzyme activity (up to 7.7-fold) in cells from the patients. Bezafibrate also diminished the production of long-chain acyl-carnitines by 90% in cells harboring moderate VLCAD deficiency. The same group also investigated the response to bezafibrate as a function of genotype in 33 VLCAD-deficient fibroblasts representing 45 different mutations. Treatment with bezafibrate resulted in a marked increase in FAO capacities, often leading to restoration of normal values, for 21 genotypes that mainly correspond to patients with the myopathic phenotype (Gobin-Limballe et al., 2007).

Situation of the research area and results by the investigator in this area The above data provided the first evidence for a possible pharmacological effect of PPAR agonists on FAO defects in humans. In the last two years, a pilot clinical trial assessing the potential beneficial effects of bezafibrate on the muscular form of CPT II deficiency has been performed in collaboration between Pitié-Salpêtrière and Necker hospitals (appel d'offre AFM 2004). Six adult patients with CPT II-deficiency received a daily 400 mg dose of bezafibrate during 6 months. Clinical tolerance of the treatment was excellent, and muscular symptoms improved in 5/6 patients with a decrease in myalgia intensity and duration. In vitro analyses were carried out on lymphocytes and skeletal muscle, sampled prior to- and at the end of the study. LCFAO in isolated muscle mitochondria was strongly induced in 6/6 patients, and this effect was shown to result from drug-induced up-regulation of CPT2 mRNA and protein levels (Djouadi et al., 2007). However the major endpoints of this study were mainly biochemical analysis, and we were not able to clearly demonstrate a decrease in the frequency of rhabdomyolysis attacks, neither an improvement of in vivo muscle metabolism.

We propose to evaluate the effect of bezafibrate on metabolism during exercise in adult patients affected with CPT II or VLCAD deficiencies. This study will be an 11-month, randomized double blind, placebo-controlled crossover trial. The trial will be conducted in two centers: Institut de Myologie, Pitié-Salpêtrière Hospital in France and Neuromuscular Research Unit, Rigshospitalet, University of Copenhagen, in Denmark. Since exercise test on cycle ergometer after stable isotopes infusion is probably the most reliable way to assess in vivo fat oxidation, this technique will be utilized as the one of two major outcomes for this study, and the main criteria for assessing the potential effect of this drug will be the fat oxidation rate during a moderate workload on cycle ergometer.

The two primary outcomes to asses the potential effect of Bezafibrate are:

• Fat oxidation and heart rate generated during physical activity on cycle ergometer at a constant workload.

We expect the fat oxidation in the patients to increase by a factor 1.7.

Secondary outcomes:

* Enzyme activity in leucocytes
* Acylcarnitine profile
* Accelerometer
* Borg score (perceived exertion)
* Number of episodes of myoglobinuria
* Daily muscle pain score (VAS)
* Daily diary of energy utilization (Bouchards questionnaire)

Material and methods:

Subjects This study will be an 9-month, randomized, double blind, placebo-controlled, crossover trial. Based on the calculation of strength in the section of statistics 22 patients, respectively 11 patients with CPT II and 11 patients with VLCAD deficiency will be included in the study:

The adult forms of CPTII and VLCAD deficiencies are very rare diseases. Twenty-five patients with CPTII deficiency and 15 patients with the myopathic form of VLCAD deficiency are currently followed in our two groups. In case that we can't include enough patients from Denmark and France, we will include patients from our collaborators in the Netherlands and Sweden. All studies will be conducted at Rigshospitalet and Pitié-Salpêtrière Hospital. Only the regularly blood samples will be outsourced to other hospitals, but the results will be faxed or mailed directly to the sponsor or investigators.

The study will be conducted on the two centers:

1. Neuromuskulær Forskningsenhed, Rigshospitalet, Danmark
2. Institut de Myologie, Pitié-Salpêtrière Hospital, Frankrig In collaboration with
3. Copenhagen Region Pharmacy, Alice Rosendahl, Marielundvej 25, Herlev, Denmark
4. Copenhagen Muscle Research Center, Rigshospitalet, Blegdamsvej 9, København Ø, Denmark
5. GCP-unit, Bispebjerg hospital, Bispebjerg Bakke 23, København NV, Denmark

The study is divided into four periods:

* First period: 1 month observation period.
* Second period: 3 months treatment with either Bezafibrate or placebo.
* Third period: 2 months wash out.
* Fourth period: 3 months treatment with either Bezafibrate or placebo (the opposite drug as in the second period).

Patients are to fill out daily scores of muscle pain (VAS score) and energy utilization (Bouchards questionnaire) during all four periods.

First period:

1. Prior to the randomizing all patients have a 1 month observation period.
2. Creatin kinase will be measured regularly in this period to define the level of muscle damage before treatment.
3. To determine a workload of 50% of maximal oxygen uptake (VO2max) for the experiment, all subjects will complete a maximal incremental cycle exercise test on a cycle ergometer in the end of this period.

Second and fourth period:

1. Subjects will be instructed to follow a standardized carbohydrate rich diet three days prior to the experiment containing 65% carbohydrate, 15% protein and 20% fat.
2. Fat oxidation study: After the 3 months observation period subjects will meet in the lab at 9.00 a.m. Two catheters will be inserted in arm veins, one in the cubital vein for stable isotope infusion and one in the distal cephalic vein for blood sampling. The subjects will receive a primed, constant rate infusion of [U-13C]-palmitate (0.0026 mg kg-1 min-1, primed by a 0.085 mg kg-1 NaH13CO3 bolus, NB! non-radioactive and non-dangerous tracers). Two hours after the start of the isotope infusion, subjects will cycle to exhaustion or for maximum 60 min. at a workload of 50-60% of VO2max as previously determined. Heart rate and the level of perceived exertion (Borg Scale) will be monitored every other minute during exercise. Blood and expired gases for isotope measurements will be collected at 10 min intervals at rest and during exercise. Expired air will be collected in a 15 L Douglas bag, and 10 ml air samples from the bags will be injected into vacutainer tubes for analyses of 13CO2 enrichment. Blood samples for acyl carnitines will be collected after 30 and 60 min. of exercise or at exhaustion, and three hours after exercise. Enzyme activity of CPT II and VLCAD will be measured on leucocytes. The above-described test will be executed both before and after each treatment period.
3. Patients will be randomized into two groups, to receive either 3 x 200mg bezafibrate or placebo in the second period and vice versa in the fourth period. Patients and all health care personal are blinded for the treatment. The randomization is carried out by the GMP-certified regional pharmacy of Copenhagen.
4. On the first trial day of these two periods patients will have blood samples taken to analyse creatin kinase, cholestrol, triglycerides, lipoproteins, total long-chain fatty acids, total carnitine, acylcarnitines, bilirubin, creatinin, aspartate amino transferase (ASAT), alanine amino transferase (ALAT), γ glutamyl transferase and alcalic phosfatase.
5. To indicate their activity level, the patients will carry an accelerometer the last fourteen days of each treatment period.

Third period:

1. Two months wash-out period.
2. Measurements of creatin kinase levels every second week.

Statistical analysis

Strength calculation:

Double blinded, randomised and crossover:

(z1-α/2 + Z1-β )2 * SD2 n ≥ _________________________ d2

Z1-α/2 = 1.96; Risk for type 1 error (α=0.05) Z1-β = 0.84; Risk for type 2 error: (1-β) = 80% SD2 = 1.25; delta palmitate oxidation in four patients with CPT II deficiency = 1.26±1.12 (Ørngreen et al, 2005) d2 = 0.87; (MIREDIF) increase in palmitate oxidation during exercise from the level of the patients with double CPT2 gene mutations to the level of the single CPT2 gene mutation subjects. (Ørngreen et al, 2005).

(1.96 + 0.84 )2 * 1.25 n ≥ _________________________ = 11 0.87

The strength calculation is based on a former study of fat oxidation in patients with CPT II deficiency. Ørngreen et al 2005 In this study we described fat oxidation of patients and carriers with respectively two and one CPT2 gene mutations compared with the fat oxidation in healthy controls. The expected effect of bezafibrate on the fat oxidation in the CPT II patients is expected to be the difference between the mean value of fat oxidation in patients with CPT II deficiency and the mean value of the fat oxidation in heterozygous carriers of one CPT2 gene mutations. The strength calculation indicates that a number of 11 subjects need to be included. The aim is to include 11 patients from respectively the groups of patients with CPT II deficiency and the groups of patients with VLCAD deficiency. If somehow it turns out that we cannot include that many patients. The two groups will be pooled into one group. This can be done because of the similarity of the two groups both in symptoms and in fat oxidation, which is one of the primary outcomes, during exercise.Ørngreen et al 2005, Ørngreen et al 2004 Missing data: As long as a patient has completed at least one treatment period, results will be included in the data. Differences between treatments in the individual will be assessed by a paired Student's t-test. A p value < 0.05 (two-tailed testing) will be considered significant.

Patients

Inclusion criteria:

1. Significant decrease in the CPT II or VLCAD activities measured in lymphocytes or fibroblasts, together with genetic verification of either CPT II deficiency or VLCAD deficiency.
2. Males and females age 18-65 years.
3. All fertile females have to have a negative pregnancy test and use anti-conceptive during the study period.

Exclusion criteria:

1. Ingestion of competitive drugs, as described in the product resume of bezafibrate.
2. Competitive disorders, evaluated by the sponsor or investigators
3. Pregnancy or lactation during the period of fibrate therapy

Safety parameters:

* CK before and every other week ± one week during treatment period.
* Hepatic enzymes (AST, ALT, γGT, alkaline phosphate), bilirubine,creatinine, cholesterol, triglycerides before treatment period, at 1 month ± one week and end of treatment period. Blood samples will be taken at local hospitals and the results will be faxed to sponsor or investigators.
* All patients will be informed to contact one of the doctors involved in case of: 1) symptoms of their disease or 2) side effects of the treatment.

Following steps are followed to ensure compliance of the patients during the treatment periods.

* Patients will be contacted weekly by mail or telephone, to ensure that the treatment is followed and that there are no symptoms of the disease or side effects of the treatment.
* In case one of the patients forget to follow the prescription of the drugs, the treatment period will be prolonged after evaluation of the sponsor or investigators.

Drugs:

In this study we use the fibrate Bezafibrate. For detailed information of effect and side effects, please see attached file with the product resume of Bezafibrate.

Randomizing and un-blinding: All drugs are delivered blinded and randomized from the pharmacy. In occurrence of life threatening or other unacceptable side effects of the treatment, a patient can be un-blinded after decision from sponsor or investigator. The randomization list will be kept by secretary Malene Kronborg Have and MD Tina Dysgaard Jeppesen in Denmark. These two persons are available 24 hours a day and are not involved in the study otherwise.

ELIGIBILITY:
Inclusion Criteria:

* CPT II or VLCAD deficiency

Exclusion Criteria:

* Competing disorders
* Liver or kidney disease
* Allergy towards fibrates
* Pregnancy and breastfeeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-10; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Fatty acid oxidation | Two years

SECONDARY OUTCOMES:
Heart rate | Two years

CONTACTS AND LOCATIONS:
Locations (1):
- Neuromusculare Research Unit, Rigshospitalet, Copenhagen, Copenhagen, Denmark

REFERENCES:
- [Background] References - Andresen BS, Olpin S, Poorthuis BJHM, Scholte HR, Vianey-Saban C, Wanders R et al. Am J Hum Genet 1999; 64: 478-494 - Bonnefont JP, Taroni F, Cavadini P, Cepanec C, Brivet M, Saudubray JM, Leroux JP, Demaugre F, (1996) Am J Hum Genet 58:971-978. - Demaugre F, Bonnefont JP, Colonna M, Cepanec C, Leroux JP, Saudubray JM. (1991) J Clin Invest 87:859-864. - DiMauro S, Melis-DiMauro PM. Science 1973;182: 929-931. - Djouadi F, Bonnefont JP, Thuillier L, Droin V, Khadom N, Munnich A, Bastin J. (2003a). Pediatr Res. 54:446-51 - Djouadi F, Bonnefont JP, Munnich A, Bastin J. (2003b). Mol Genet Metab.;78:112-8. - Djouadi F, Aubey F, Schlemmer D, Ruiter JPN, Wanders RJA, Strauss AW et al. Hum Mol Genet 2005; 18: 2495-2703 - Djouadi F, Aubey F, Schlemmer D, Ruiter JPN, Wanders RJA, Strauss AW et al. Hum Mol Genet 2005; 14:2695-2703. - Djouadi F, Aubey F, Schlemmer D, Gobin S, Laforet P, Wanders RJA, et al. J Inherit Metab Dis 2006; 29: 341-342. - Djouadi F, Bastin J, Laforêt P, Aubey F, Mogenet A, Romano S et al. ASHG 57th Annual meeting (2007). - Johansen K. Basal Sundhedsvidenskabelig statistik. Munksgaard, Denmark 2002 1st edition. - Lemberger T, Desvergne B, Wahli W (1996) Annu. Rev. Cell. Dev. Biol. 12:335-363. - Ørngreen MC, Ejstrup R, Vissing J. Neurology 2003; 61:559-561. - Ørngreen MC, Nørgaard MG, Sacchetti M, van Engelen BGM, Vissing J. Ann Neurol. 2004; 56:279-282. - Ørngreen MC, Dunø M, Ejstrup R, Christensen E, Schwartz M, Sacchetti M, Vissing J. Ann Neurol. 2005; 57:60-66. - Ørngreen MC, Schelhaas HJ, Jeppesen TD, Akman HO, Wevers RA, Andersen ST, Ter Laak HJ, van Diggelen OP, DiMauro S, Vissing J. INeurology, 2008;70(20):1876-82. - Roe CR, Sweetman L, Roe DS, David F, Brunengraber H. J Clin Invest 2002; 110: 259-269. - Vianey-Saban C, Divry P, Brivet M, Nada M, Zabot M-T, Mathieu M et al. Clin Chim Acta 1998; 269: 43-62.